CLINICAL TRIAL: NCT04648670
Title: Cognitive Stimulation Program in Elderly With Normal Cognition: a Randomized Controlled Trial
Brief Title: Cognitive Stimulation Program in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Isabel Gómez-Soria, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Randomized Controlled Trial; Occupational Therapy; Aging; Cognitive Change

STUDY DESIGN:
Intervention Model Description: An intervention group and a control group with the same characteristics are included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group intervention (Experimental): The experimental group consists of 101 participants have been subdivided into two groups of 25/26 that perform the same intervention but on a different day of the week.
  The two subgroups have received 10 sessions of 45 minutes/week during 10 weeks. Each session included four parts: (a) Reality orientation therapy, (b) activities related to memory, orientation, language, praxis, gnosis, calculation, perception, reasoning, visual attention, and executive functions, (c) individual practical exercises and (d) correction of the practical exercises.
  .
  Interventions: Behavioral: Cognitive stimulation
- Group Control (No Intervention): The control group consists of 100 participants. The no intervention group did not receive any type of intervention

INTERVENTIONS:
Behavioral: Cognitive stimulation — The intervention was applied to the experimental group and consisted in 10 sessions of 45 minutes/week during 10 weeks. Each session included four parts: (a) Reality orientation therapy, (b) activities related to memory, orientation, language, praxis, gnosis, calculation, perception, reasoning, visual attention, and executive functions, (c) individual practical exercises and (d) correction of the practical exercises..
  Arms: Group intervention

SUMMARY:
The participants who carry out our cognitive stimulation program maintain and / or improve their score of the 35-point Spanish version of 35 points of Mini-mental State of Folstein; Mini-exam Cognoscitive of Lobo

DETAILED DESCRIPTION:
The aim of our research is to evaluate the effect of a cognitive stimulation program in older adults aged 65 or over The intervention was carried out at the Foundation of Zaragoza (Spain), consisting of 10 sessions of 45 minutes/week during 10 weeks.with normal cognition and compare it, in the short, medium and long term, with the evolution of other people, with the same characteristics and for which this intervention has not been carried out.

The significant increase in the number of people over 65 years of age in relation to the total population suggests a significant increase in age-related pathologies. Prevention is essential to avoid cognitive aging and preserve higher mental functions.

From an economic perspective, it is estimated that people with mild cognitive impairment produce 16% more spending than those with normal cognition.

Cognitive stimulation is a low-cost non-pharmacological treatment that has shown its benefits in the preservation of cognitive aspects based on the brain plasticity it generates.

Our research is based on cognitive stimulation using the yellow and Orange Mental Activation notebooks, levels that correspond to the scores of Lobo's cognitive Mini-test. The book consists of 4 practical exercises that work on 10 cognitive aspects (memory, orientation, language, praxis, gnosis, calculation, perception, reasoning, attention and programming); in total 40 exercises. The models on which the laptop is based are the cognitive model and the human occupation model.

In the Health Center San José Norte-Centro of Zaragoza (Spain), assessments were made to 416 volunteer candidates, of which 215 were excluded for not meeting the inclusion criteria; being a total of 201participants that have been part of the randomized controlled trial. Of the 201 participants; 101 have carried out the intervention as an intervention group and 100 as the control group. The control group did not perform any type of intervention.

The intervention was carried out at the Foundation of Zaragoza (Spain), consisting of 10 sessions of 45 minutes/week during 10 weeks.

The conceptual framework of this intervention is formed by the framework for practice of Occupational Therapy, the cognitive model and the human occupation model of Gary Kielhofner .

To homogenize both the assessments and the intervention, a standardized training was carried out for the occupational therapists who carried them out and consisted of a theoretical part and a practical part of 10 hours each.

The study began in December 2011, obtained the authorization of the Directorate of Primary Care of the Zaragoza II Sector and the approval of the project by the Research Ethics Committee of the Government of Aragón (CEICA). This study has followed the ethical standards recognized by the Declaration of Helsinki. The initial assessments began this month. The necessary sample size was reached in October 2012 and, from that moment on, randomization and intervention with the selected participants was carried out. Three other assessments were made, both for the intervention group and for the control group, immediately after the intervention, six months and one year after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Older adults (age ≥ 65)
* Older people with an MEC between: 28-35 points with or without psychiatric pathology (depression, anxiety)
* Non-Institutionalized People.
* Older people with a Lawton index greater than or equal to 3.

Exclusion Criteria:

* People who have received some type of cognitive stimulation therapy in the last year, that is, people who attend memory or mental activation workshops (in the major centers of the Zaragoza City Council, elderly associations, women's associations, etc. .).
* People who present values of more than 6 points, in the abbreviated Goldberg anxiety scale and also in the Yesavage depression scale, score more than 12/15, due to presenting intense symptoms, which made it difficult to carry out the intervention.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 201 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2012-10-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
The Spanish versions of the Mini-Mental State Examination (MEC-35) | baseline and change in 1 week, 6 months, baseline and 12 moths
  It is a reliable and used instrument for the evaluation of cognitive impairment. It meets criteria of "feasibility", "content validity", "procedural" and "construction". Test-retest reliability: weighted kappa = 0.667, sensitivity = 89.8%, and specificity = 83.9%; with the cutoff point 23/24. A score of 28 is considered the lower limit of normal performance in adult population; scores equal or less than 27 would denote cognitive deficits.

SECONDARY OUTCOMES:
Set Test | baseline and change in 1 week, 6 months, baseline and 12 moths
  The set-test was first introduced by Isaacs in 1972, and proposed as an aid in the diagnosis of dementia in the elderly population by Isaacs and Kennie in 1973. It explores verbal fluency, category naming and semantic memory. The collection of information is through a hetero-administered questionnaire. Adapted and validated by Dr. Pascual. It measures the verbal fluency of a categorical type, by asking the subject to cite up to a maximum of ten responses from each of the following categories: colors, animals, fruits and city. There is extensive experience in the use of this scale in our country. It is an option in illiterate people, with sensory impairments or when the consultation time is a conditioning factor. It has a sensitivity of 87% and a specificity of 67%, with a misclassification rate of 24% .The cut-off point to detect dementia: -In adults: Equal to or less than 29 -In older than 65 years: Equal to or less than 27
The Barthel Index (Barthel) | baseline and change in 1 week, 6 months, baseline and 12 moths
  Developed by Mahoney & Barthel (1965), assesses the level of independence in ten Basic Activities of Daily Living (BADLs) and is an indicator of skills for people with reduced mobility. Its internal consistency is 0.89-0.92; obtains intra- observer reliability with kappa indexes between 0.47 to 1.0. Values the ability to perform ten BADLs: feeding, bathing, dressing, grooming, bowel control, bladder control, toilet use, transfers chair-bed, mobility and stairs use. A score is assigned to each item (0, 5, 10, 15) as a function of time and help needed. The final score varies from 0 (completely dependent) to 100 (completely independent). Above 60 points there is a high probability of continuing to live in the community.
The scale of Lawton & Brody (Lawton) | baseline and change in 1 week, 6 months, baseline and 12 moths
  Assesses the degree of autonomy in eight Instrumental Activity Daily Livings (IADLs) necessary for living independently in the community. Its reliability is = 0.85 sensitivity = 0.57 and specificity = 0.92. In a study in Spanish population the internal consistency was 0.94; Regarding the convergent validity all the correlation coefficients were higher than 0.40. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men (historically, for men, the areas of food preparation, housekeeping, laundering are excluded).
The Goldberg questionnaire (EADG) | baseline and change in 1 week, 6 months, baseline and 12 moths
  Evaluates the mood referred to anxiety and depression. The original questionnaire was developed by Goldberg and consisted of 18 items. Consists of two sub-scales, one of anxiety and other of depression. The last 5 questions of the EADG are only formulated if there are positive answers to the first 4 questions, which are obligatory. The higher the number, the more severe your depression is likely to be. Of all the cutoff points, the most suitable result for the sub-scale of anxiety is 4 points and for the sub-scale of depression is 2 point. The Spanish version of EADG has demonstrated its reliability and validity in the field of Primary Care; with a sensitivity of 83.1%, a specificity of 81.8%, a misclassified index of 17.7% and a positive predictive value of 95.3% .
  The investigators used the sub-scale of anxiety; its overall specificity = 91% and its sensitivity = 86%
The abbreviated Yesavage depression scale (GDS-15) | baseline and change in 1 week, 6 months, baseline and 12 moths
  Evaluates the mood referred to depression. The first version consisted of 30 items . Subsequently, abbreviated version (GDS-15) was published with 15 questions; for use in older people living in the community. For cut-off point 4/5 the sensitivity rates vary between 92.7% and 97.0%, the specificity between 54.8% and 65.2%; the positive predictive value between 69.6% and 82.6% and the negative between 83.3% and 94.4%.

REFERENCES:
- [Background] Lobo A, Saz P, Marcos G, Dia JL, de la Camara C, Ventura T, Morales Asin F, Fernando Pascual L, Montanes JA, Aznar S. [Revalidation and standardization of the cognition mini-exam (first Spanish version of the Mini-Mental Status Examination) in the general geriatric population]. Med Clin (Barc). 1999 Jun 5;112(20):767-74. Spanish. PMID 10422057
- [Background] Goldberg D, Bridges K, Duncan-Jones P, Grayson D. Detecting anxiety and depression in general medical settings. BMJ. 1988 Oct 8;297(6653):897-9. doi: 10.1136/bmj.297.6653.897. PMID 3140969
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Background] Pascual Millan LF, Martinez Quinones JV, Modrego Pardo P, Mostacero Miguel E, Lopez del Val J, Morales Asin F. [The set-test for diagnosis of dementia]. Neurologia. 1990 Mar;5(3):82-5. Spanish. PMID 2361045
- [Background] Lee SW, Taylor R, Kielhofner G, Fisher G. Theory use in practice: a national survey of therapists who use the Model of Human Occupation. Am J Occup Ther. 2008 Jan-Feb;62(1):106-17. doi: 10.5014/ajot.62.1.106. PMID 18254437
- [Background] Vinyoles Bargallo E, Vila Domenech J, Argimon Pallas JM, Espinas Boquet J, Abos Pueyo T, Limon Ramirez E; Los investigadores del proyecto Cuido 1*. [Concordance among Mini-Examen Cognoscitivo and Mini-Mental State Examination in cognitive impairment screening]. Aten Primaria. 2002 Jun 15;30(1):5-13. doi: 10.1016/s0212-6567(02)78956-7. Spanish. PMID 12106573
- [Background] Hanninen T, Koivisto K, Reinikainen KJ, Helkala EL, Soininen H, Mykkanen L, Laakso M, Riekkinen PJ. Prevalence of ageing-associated cognitive decline in an elderly population. Age Ageing. 1996 May;25(3):201-5. doi: 10.1093/ageing/25.3.201. PMID 8670552
- [Background] Novoa AM, Juarez O, Nebot M. [Review of the effectiveness of cognitive interventions in preventing cognitive deterioration in healthy elderly individuals]. Gac Sanit. 2008 Sep-Oct;22(5):474-82. doi: 10.1157/13126930. Spanish. PMID 19000530
- [Background] Duara R, Loewenstein DA, Greig M, Acevedo A, Potter E, Appel J, Raj A, Schinka J, Schofield E, Barker W, Wu Y, Potter H. Reliability and validity of an algorithm for the diagnosis of normal cognition, mild cognitive impairment, and dementia: implications for multicenter research studies. Am J Geriatr Psychiatry. 2010 Apr;18(4):363-70. doi: 10.1097/jgp.0b013e3181c534a0. PMID 20306566
- [Background] Pusswald G, Tropper E, Kryspin-Exner I, Moser D, Klug S, Auff E, Dal-Bianco P, Lehrner J. Health-Related Quality of Life in Patients with Subjective Cognitive Decline and Mild Cognitive Impairment and its Relation to Activities of Daily Living. J Alzheimers Dis. 2015;47(2):479-86. doi: 10.3233/JAD-150284. PMID 26401569
- [Derived] Gomez-Soria I, Ferreira C, Olivan-Blazquez B, Aguilar-Latorre A, Calatayud E. Effects of cognitive stimulation program on cognition and mood in older adults, stratified by cognitive levels: A randomized controlled trial. Arch Gerontol Geriatr. 2023 Jul;110:104984. doi: 10.1016/j.archger.2023.104984. Epub 2023 Mar 4. PMID 36921506
- [Derived] Gomez-Soria I, Cuenca-Zaldivar JN, Rodriguez-Roca B, Subiron-Valera AB, Salavera C, Marcen-Roman Y, Andrade-Gomez E, Calatayud E. Cognitive Effects of a Cognitive Stimulation Programme on Trained Domains in Older Adults with Subjective Memory Complaints: Randomised Controlled Trial. Int J Environ Res Public Health. 2023 Feb 18;20(4):3636. doi: 10.3390/ijerph20043636. PMID 36834329